CLINICAL TRIAL: NCT05017870
Title: A Randomized, Double-blinded, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristic of KSR-001 in Healthy Male Volunteers
Brief Title: [KSR-001-P01]Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristic of KSR-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kukje Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSR-001-P01
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KSR-001-01 (Experimental): Participants received KSR-001-01 for 6 days.
  Interventions: Drug: KSR-001
- KSR-001-02 (Experimental): Participants received KSR-001-02 for 6 days.
  Interventions: Drug: KSR-001-02
- KSR-001-03 (Experimental): Participants received KSR-001-03 for 6 days.
  Interventions: Drug: KSR-001-03
- KSR-001-04 (Placebo Comparator): Participants received KSR-001-04 for 6 days.
  Interventions: Drug: KSR-004

INTERVENTIONS:
Drug: KSR-001 — (0 day) eye drops received one drop to both eyes once a day (1~5 day) eyedrops recieved one drop to both eyes four times a day
  Other Names: KSR-001-01
  Arms: KSR-001-01
Drug: KSR-004 — (0 day) eye drops received one drop to both eyes once a day (1~5 day) eyedrops recieved one drop to both eyes four times a day
  Arms: KSR-001-04
Drug: KSR-001-02 — KSR-001-02
  Arms: KSR-001-02
Drug: KSR-001-03 — KSR-001-03
  Arms: KSR-001-03

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetic characteristic of KSR-001.

DETAILED DESCRIPTION:
After single dose, safety and local tolerability were confirmed and repeated test was conducted according to the investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 19 and 45 years of age inclusive, at the time of signing the informed consent.
2. Body weight >= 50 kilogram and ideal body weight within the range ±20%.
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. A subject who has symptoms of suspected acute disease at the time of screening.
2. Subjects with a history of abnormal digestive organ, kidney, respiratory, neuroendocrine, cardiovascular, hemato-oncology, urinary, musculoskeletal, immune, the nose and ears, psychiatry, stomach system.
3. A subject determined to be unsuitable as a subject through a physical examined during screening.
4. A subject who is determined to be unsuitable as a subject through an ophthalmologic examination performed during screening.
5. A subject with a history of ophthalmic surgery, trauma and chronic diseases.
6. A subject who has acute or chronic eye disease requiring the use of local eye drops at the time of screening.
7. Subjects who need to wear contact lenses during clinical trial period.
8. A subject with clinically significant allergic disease.
9. A subject with a history of drug abuse.
10. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator contraindicates their participation.
11. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days of the biological effect of the investigational product (whichever is longer).
12. A subject who takes drugs that induce and inhibit drug metabolises such as barbital medicines within one month before the administration of clinical trial drugs.
13. A subject who donates blood to the whole blood within 60 days before the administration of a clinical trial drug or a person who donates blood to the component within 20 days before the administration of a clinical trial drug.
14. A subject who has taken a specialty drug or herbal medicine within 14 days of administration of a clinical trial drug or a general medicine or vitamin formulation within 7 days.
15. A subject who can not continually ingest caffeine or ingest caffeine-containing foods during the period from 24 hours to discharge from hospital.
16. A subject who can not drink alcohol continuously or during the period from 24 hours to discharge from hospital.
17. A subject who can not smoke excessively or quit smoking during the period from 24 hours to discharge from hospital.
18. A subject who investigator that a tester is unsuitable for participating in clinical trials due to other reasons.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 6 days
  Pharmacokinetic Characteristics
Tmax | 6 days
  Pharmacokinetic Characteristics
t1/2 | 6 days
  Pharmacokinetic Characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Kukje Pharma, Seongnam-si, South Korea